CLINICAL TRIAL: NCT02483208
Title: Single Dose, Open-label, Randomized, Crossover Study in Subjects With Severe Hemophilia A Comparing Pharmacokinetic Parameters for BAY81-8973 and Advate
Brief Title: Single Dose Study in Subjects With Severe Hemophilia A Comparing Pharmacokinetic Parameters for BAY81-8973 and Advate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17608; 2014-005173-36 (EudraCT Number)
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BAY81-8973 (Experimental): BAY81-8973 infusion to analyze pharmacokinetics
  Interventions: Drug: BAY81-8973
- Advate (Other): Advate infusion to analyze pharmacokinetics.
  Interventions: Drug: Advate

INTERVENTIONS:
Drug: BAY81-8973 — BAY81-8973 infusion to analyze pharmacokinetics
  Arms: BAY81-8973
Drug: Advate — Advate infusion to analyze pharmacokinetics.
  Arms: Advate

SUMMARY:
The purpose of this study is to compare the pharmacokinetics of BAY81-8973 and Advate after intravenous administration.

ELIGIBILITY:
Inclusion Criteria:

* Males, age 18 to 65 years

  * Subjects with Severe hemophilia A with a documented plasma FVIII level of <1%
  * ≥ 150 exposure days with FVIII concentrate(s) as supported by medical records

Exclusion Criteria:

* Evidence of current or past inhibitor antibody

  * History of any congenital or acquired coagulation disorders other than hemophilia A
  * Platelet count <75,000/mm3
  * Abnormal renal function (serum creatinine >2 times the upper limit of the normal [ULN] range)
  * Active liver disease verified by medical history or persistently elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 times the ULN or severe liver disease as evidenced by, but not limited to any of the following: International Normalized Ratio (INR) >1.4, hypoalbuminemia, portal vein hypertension including presence of otherwise unexplained splenomegaly and history of esophageal varices.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
AUC(0-tlast) | Pre-Dose, 0.25, 0.5, 1, 3, 6, 8, 24, 30, 48 hours after treatment
  Area under the blood concentration vs time curve from zero to the last data point > lower limit of quantification

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Sofia, Bulgaria

REFERENCES:
- [Derived] Shah A, Solms A, Garmann D, Katterle Y, Avramova V, Simeonov S, Lissitchkov T. Improved Pharmacokinetics with BAY 81-8973 Versus Antihemophilic Factor (Recombinant) Plasma/Albumin-Free Method: A Randomized Pharmacokinetic Study in Patients with Severe Hemophilia A. Clin Pharmacokinet. 2017 Sep;56(9):1045-1055. doi: 10.1007/s40262-016-0492-2. PMID 28005225